CLINICAL TRIAL: NCT06432816
Title: Efficacy of Nano-Pso Therapy Compared to Placebo in the Control of Vasomotor Symptomatology in Early Menopause
Brief Title: Efficacy of Nano-Pso Therapy in Menopause
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Distribuidora Biolife SA de CV (Industry)
Responsible Party: Principal Investigator, Dra Araceli Espinosa Guerrero, DRA. Araceli Espinosa Guerrero, Distribuidora Biolife SA de CV
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMI-09-23
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Menopause; Vasomotor; Syndrome
MeSH Terms: conditions — Syndrome | interventions — Nano-PSO; Nanotechnology

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, analytical and longitudinal study. A sample calculation was made with a therapeutic efficiency of 30% in vasomotor syndrome, with a result of 210 participants, divided into 3 institutions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treatments were received, previously labeled and randomly drawn by the sponsor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NANO-PSO (Active Comparator): NANO-PSO or Pomegranate seed oil with nanotechnology, capsules with a net content of 640 mg with a dosage indicated by sponsor of 2 capsules in fast
  Interventions: Dietary Supplement: NANO-PSO
- PLACEBO (Placebo Comparator): - Placebo physically identical to NANO-PSO capsules: Soft gelatin capsules 640 mg edible oil 35for PLACEBO being the following information: Oil edible, oval shape, 640 mg.
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: NANO-PSO — NANO-PSO or Oil of pomegranate seed with nanotechnology, they are capsules with a net content of 640 mg with a dosage indicated by sponsor of 2 capsules in fast
  Other Names: Oil of pomegranate seed with nanotechnology
  Arms: NANO-PSO
Other: PLACEBO — Placebo physically identical to NANO-PSO capsules:
  Soft gelatin capsules 640 mg edible oil 35for PLACEBO Oil edible, oval shape, 640 mg.
  Arms: PLACEBO

SUMMARY:
Vasomotor syndrome is prevalent in 85% of postmenopausal women, hormone therapy in menopause is first-line therapy, but 38% of patients have some contraindication for its use. The medications indicated in this population presents adverse reactions, such as dryness of the mucous membranes, and insomnia in patients, and triggers to abandoned treatment due to poor response to the drug. Aligned with the safety of patients, we wish to test pomegranate seed oil with nanotechnology (NANOPSO), which has been reported to have positive results at a central level, due to its antioxidant effect, which could impact women in climacteric in a positive way. The study involves the participation of 90 patients divided into two groups, where placebo or Nano-PSO will be administered for 60 days, with a total follow-up of 120 days. It is established that patients must not have received previous treatments for menopausal symptoms. Therefore, it is expected that therapy with NANO-PSO compared to placebo will be more effective in controlling vasomotor symptoms in early menopause after 6 months of treatment evaluated by the MRS scale.

DETAILED DESCRIPTION:
The menopausal transition in women marks the end of female reproductive capacity and is associated with an estrogenic hormonal imbalance that begins to be noticeable around the fifth decade of life. This process, also known as climacteric, involves the transition from an active to an inactive reproductive stage, and can last for several years before menopause, which is defined as the last menstruation .

During the climacteric, the reduction of estrogen triggers clinical signs and symptoms that affect various systems of the body, such as the central nervous system, the cardio-metabolic system, the musculoskeletal system, and sexual function. Vasomotor symptoms, such as hot flashes, are common manifestations at this stage and affect approximately 75-80% of women in the transition to menopause, with an intensity ranging from moderate to severe in most cases. These symptoms can have a negative impact on quality of life, affecting sleep, functional capacity and work attendance .

Menopausal hormone therapy (MHT) with estrogens and progesterone is the first line of treatment for vasomotor symptoms in menopause. However, some women cannot or prefer not to use MHT due to its adverse effects, which has led to the development of second-line therapies, such as selective serotonin reuptake inhibitors, gabapentinoids, clonidine, and oxybutynin. These non-hormonal therapies may also have minor side effects that may lead to discontinuation of treatment.

In the search for therapeutic alternatives with fewer adverse effects, compounds such as punic acid (omega 5) and its metabolites, such as conjugated linoleic acid, have been investigated. Nanoemulsified pomegranate seed oil (omega 5) has been shown to be a compound with high antioxidant capacity and neuroprotective effects, making it a promising option for the management of symptoms associated with menopause, especially those related to alterations at the level of the menopause. central. Preliminary studies have shown encouraging results in animal models and initial clinical trials, suggesting the need for additional research in specific populations, such as menopausal women.

GENERAL OBJECTIVE

Compare 6-month NANO-PSO therapy versus placebo in the control of vasomotor symptoms in early menopause, assessed via the Menopause Rating Scale.

SPECIFIC OBJECTIVES

* Describe the sociodemographic and clinical characteristics of the Study population.
* Analyze vasomotor symptoms in menopausal patients at baseline with the MRS scale.
* Compare vasomotor symptoms with the use of NANO-PSO vs. Placebo
* Compare the percentage of treatment response regarding vasomotor symptoms with the use of nano pso vs placebo at 3 and 6 months.

Population study Patients who come first class. outpatient climacteric consultation that presents with early menopause and MRS scale > 15 points without treatment.

With a sample convenience, the aim is to recruit 45 patients per group with a total of 90 patients. Intervention by compounds - Leading to treatment of NANO-PSO or Oil of pomegranate seed with nanotechnology, they are capsules with a net content of 640 mg with a dosage indicated by sponsor of 2 capsules in fast

- Placebo physically identical to NANO-PSO capsules: Soft gelatin capsules 640 mg edible oil 35for PLACEBO being the following information: Oil edible, oval shape, 640 mg.

ELIGIBILITY:
Inclusion Criteria:

* In perimenopause with vasomotor syndrome and score greater than 15 points staged with the MRS scale
* They agree to participate and sign the consent informed.
* Without prior treatment to relieve the symptoms of menopause.

Exclusion Criteria:

* - With pharmacological and/or hormonal therapy prescribed for menopause symptoms.
* With psychiatric pathologies such as anxiety and depression.
* Hysterectomized patients or patients with induced menopause surgically early.
* Smoking
* Malnutrition or low weight determined by a BMI ≤ 18.5Kg/m2

Elimination criteria.

* Who do not attend follow-up to provide their treatment the 1, 2, 3 and 4 months for application of the MRS scale
* That they leave the study voluntarily.
* Who present any serious adverse effect to the drug.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
MENOPAUSE RATING SCALE | 1 BASELINE EVALUATION WILL BE CARRIED OUT AFTER 3 AND SIX MONTHS.
  THE MRS IS A SCALE TO IDENTIFY THE FREQUENCY AND INTENSITY OF MENOPAUSE SYMPTOMS
FSH HORMONE | 1 BASELINE EVALUATION WILL BE CARRIED OUT AFTER 3 AND SIX MONTHS.
  Follicle-stimulating hormone (FSH) is a pituitary hormone that regulates the reproductive cycle, helps control the menstrual cycle and the production of eggs in the ovaries.
PITTSBURG SCALE | 1 BASELINE EVALUATION WILL BE CARRIED OUT AFTER 3 AND SIX MONTHS.
  The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire commonly used to evaluate sleep quality in adults. Created by the Department of Psychiatry at the University of Pittsburgh in 1988, the PSQI addresses both qualitative and quantitative aspects of sleep experienced during the month prior to its administration.
STRAW+10 | 1 BASELINE EVALUATION WILL BE CARRIED OUT AFTER 3 AND SIX MONTHS.
  The STRAW+10 system is a clinical and objective way to stage patients transitioning to menopause.

SECONDARY OUTCOMES:
PHQ-9 | 1 BASELINE EVALUATION WILL BE CARRIED OUT AFTER 3 AND SIX MONTHS.
  The PHQ-9 is a nine-item self-report measure that assesses the presence of depressive symptoms based on DSM-IV criteria.
ESTRADIOL | EVALUATION WILL BE CARRIED OUT AFTER SIX MONTHS.
  Estradiol is a female sex hormone that regulates many processes in the body in the reproductive age, its evaluation will only be a control.

CONTACTS AND LOCATIONS:
Overall Officials: ARACELI ESPINOSA GUERREO, Principal Investigator — Maternal and child institute of the State of Mexico
Locations (1):
- Maternal and Child Institute of the State of Mexico, Toluca, State of Mexico, Mexico

REFERENCES:
- [Background] El Khoudary SR, McClure CK, VoPham T, Karvonen-Gutierrez CA, Sternfeld B, Cauley JA, Khalil N, Sutton-Tyrrell K. Longitudinal assessment of the menopausal transition, endogenous sex hormones, and perception of physical functioning: the Study of Women's Health Across the Nation. J Gerontol A Biol Sci Med Sci. 2014 Aug;69(8):1011-7. doi: 10.1093/gerona/glt285. Epub 2014 Jan 24. PMID 24465026
- [Background] Monteleone P, Mascagni G, Giannini A, Genazzani AR, Simoncini T. Symptoms of menopause - global prevalence, physiology and implications. Nat Rev Endocrinol. 2018 Apr;14(4):199-215. doi: 10.1038/nrendo.2017.180. Epub 2018 Feb 2. PMID 29393299
- [Background] Avis NE, Crawford SL, Green R. Vasomotor Symptoms Across the Menopause Transition: Differences Among Women. Obstet Gynecol Clin North Am. 2018 Dec;45(4):629-640. doi: 10.1016/j.ogc.2018.07.005. Epub 2018 Oct 25. PMID 30401547
- [Background] Kim MJ, Yim G, Park HY. Vasomotor and physical menopausal symptoms are associated with sleep quality. PLoS One. 2018 Feb 20;13(2):e0192934. doi: 10.1371/journal.pone.0192934. eCollection 2018. PMID 29462162
- [Background] Petrou P, Ginzberg A, Binyamin O, Karussis D. Beneficial effects of a nano formulation of pomegranate seed oil, GranaGard, on the cognitive function of multiple sclerosis patients. Mult Scler Relat Disord. 2021 Sep;54:103103. doi: 10.1016/j.msard.2021.103103. Epub 2021 Jun 27. PMID 34243101
- [Background] Auerbach L, Rakus J, Bauer C, Gerner C, Ullmann R, Wimmer H, Huber J. Pomegranate seed oil in women with menopausal symptoms: a prospective randomized, placebo-controlled, double-blinded trial. Menopause. 2012 Apr;19(4):426-32. doi: 10.1097/gme.0b013e3182345b2f. PMID 22240636
- [Background] Mori-Okamoto J, Otawara-Hamamoto Y, Yamato H, Yoshimura H. Pomegranate extract improves a depressive state and bone properties in menopausal syndrome model ovariectomized mice. J Ethnopharmacol. 2004 May;92(1):93-101. doi: 10.1016/j.jep.2004.02.006. PMID 15099854
- [Background] Valdes-Sustaita B, Estrada-Camarena E, Gonzalez-Trujano ME, Lopez-Rubalcava C. Estrogen receptors-beta and serotonin mediate the antidepressant-like effect of an aqueous extract of pomegranate in ovariectomized rats. Neurochem Int. 2021 Jan;142:104904. doi: 10.1016/j.neuint.2020.104904. Epub 2020 Nov 18. PMID 33220387
- [Background] Adel-Mehraban MS, Tansaz M, Mohammadi M, Yavari M. Effects of pomegranate supplement on menopausal symptoms and quality of life in menopausal women: A double-blind randomized placebo-controlled trial. Complement Ther Clin Pract. 2022 Feb;46:101544. doi: 10.1016/j.ctcp.2022.101544. Epub 2022 Feb 2. PMID 35134697
- [Background] Kim JH, Kim YJ, Park Y. Conjugated Linoleic Acid and Postmenopausal Women's Health. J Food Sci. 2015 Jun;80(6):R1137-43. doi: 10.1111/1750-3841.12905. Epub 2015 May 11. PMID 25962640
- [Background] Posadzki P, Lee MS, Moon TW, Choi TY, Park TY, Ernst E. Prevalence of complementary and alternative medicine (CAM) use by menopausal women: a systematic review of surveys. Maturitas. 2013 May;75(1):34-43. doi: 10.1016/j.maturitas.2013.02.005. Epub 2013 Mar 14. PMID 23497959